CLINICAL TRIAL: NCT02681341
Title: Vascular Post Market Review
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 015-236
Record Dates: First submitted 2016-01-22; First posted 2016-02-12 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Carotid Endarterectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to confirm that properties of CardioCel provide operative benefit to surgeons when compared to Dacron, CorMatrix, and all other bovine pericardium not treated with proprietary ADAPT engineering.

DETAILED DESCRIPTION:
ENDPOINTS

1. OR experience: suturability, handling, hemostasis, compliance to recipient vessel, blood loss, OR time.
2. In-hospital survival
3. MAE (Stroke, MI, death)
4. 1 Month duplex US scan
5. 6 month duplex US scan

Secondary Efficacy Endpoints

1. Less than 50% stenosis at 6 months (PSV <150 cm/s)

Safety Endpoint

Incidence of CardioCel related Major Adverse Cardiac Events (MACE) at 6 months, defined for this study as:

* Structural CardioCel failure - aneurysm/dilation
* Vasculitis
* Leak or pseudoaneurysm
* Dehiscence
* Thromboembolism
* Thrombosis
* Haemolysis
* Reoperation and explant

Review endpoints at 6 months to confirm results meet the expectations of the Principal Investigator.

BACKGROUND

Rationale for Study:

CardioCel's unique strength, pliability, resistance to degradation and calcification make it a promising alternative to synthetic fabrics or other xenographic materials incompletely decellularized or detoxified (aldehyde removal).

Device Description:

Tissue-engineered CardioCel pericardium is manufactured from bovine spongiform encephalopathy-free pericardium (37). Manufacturing consists of several tissue-engineering processes, which include steps to remove lipids, cells and cell remnants, nucleic acids (DNA, RNA) and Gal epitopes. In addition, cross-linking is achieved with an ultra-low engineered glutaraldehyde concentration to minimise glutaraldehyde cytotoxicity levels (Admedus Ltd. proprietary). Cytotoxicity is further reduced by the ADAPT® anti-calcification process and a non-glutaraldehyde sterilisation and storage solution.

CardioCel is US FDA cleared for the repair of cardiac and vascular defects, including intra-cardiac defects; septal defects, valve and annulus repair, great vessel reconstruction, peripheral vascular reconstruction, suture line buttressing and pericardial closure.

STUDY DESIGN This is a prospective, non-randomized, single arm study.

SCHEDULE OF ASSESSMENTS/DATA COLLECTION

ENROLLMENT:

10 subjects to be enrolled per site

DURATION OF ENROLLMENT:

Patients will be followed for 6 months after CEA procedure.

SCREENING A pre-screening procedure may be performed to determine whether the patient meets the inclusion/exclusion eligibility selection criteria. A pre-screened patient will be asked to sign the informed consent form before any study-specific tests or procedures are performed. Subject screening numbers will be assigned at this visit and subjects will be evaluated for eligibility criteria.

BASELINE Informed consent will be obtained from all subjects who are potential trial candidates prior to commencement of any study related procedures.

The following baseline data will be collected for all subjects prior to procedure:

* Patient demographics
* Standard of care Physical Examination
* Vital Signs (Blood pressure and heart rate only)
* Medical history (for cardiovascular risk factors)
* Standard of care Clinical Lab tests
* Final confirmation of Inclusion/Exclusion Criteria

IMPLANT PROCEDURE Patients will undergo a CEA with patch arterioplasty. Patients will be managed according to standard pre-operative, operative, and postoperative care.

The following OR Experience data will be collected for all subjects:

* Suturability
* Handling
* Hemostasis
* Compliance to recipient vessel
* Blood loss
* OR time
* In-hospital survival
* MAE (Stroke, MI, death)

FOLLOW-UP VISITS Patients will return for follow-up visits that will include a carotid duplex ultrasound at 1 and 6 months. Follow-up visits may also include a physical examination and adverse event review.

The following follow-up data will be collected for all subjects:

* Standard of care physical examination
* 1 Month duplex US scan- Duplex US scanning for velocity, calibre, occlusion/lesion status
* 6 month duplex US scan- Duplex US scanning for velocity, calibre, occlusion/lesion status
* MAE (Stroke, MI, death) and AE review at each visit

STATISTICAL ANALYSIS & DATA MANAGEMENT:

Principal Investigator plans to follow patients for 6 months and create report (white paper) on OR experiences and 6 month follow-up. The study is a direct observation of 6 month follow-up for patients undergoing CEA with patch arterioplasty. No control group is included in the study, and no comparative analysis is planned.

DATA MONITORING Internal monitoring will be conducted periodically. CRF's, source documents, informed consent forms, and study deviations will be included; these findings will be reported to the PI. Deviations will be documented and reported according to IRB policy. Regulatory documents will be audited by the Baylor Research Institute Department of Research Compliance upon request.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for carotid endarterectomy (CEA) with patch arterioplasty
* Expected lifespan of over 24 months
* Age over 18 years

Exclusion Criteria:

* Revision of previous CEA arterioplasty
* Active infection
* Cerebral ischemic event (completed stroke) within 30 days of planned surgery
* Pregnant or breastfeeding
* Concomitant surgical or endovascular procedure being performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing a carotid endarterectomy with patch arterioplasty
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
6 Month Duplex US Report to Measure Material Quality | Up to 6 months post CEA
  The 6 month duplex US report will measure peak velocity and flow through the repaired carotid artery, caliber, and occlusion/lesion status as per normal parameters used in post-CEA scans.

SECONDARY OUTCOMES:
OR Data and Surgeon Feedback During the Procedure | procedure
  The OR data from the procedure including blood loss and how long it took to achieve hemostasis in addition to surgeon feedback on bleeding, handling, and suturing of the material will be collected on a source worksheet.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Gable, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- The Heart Hospital Baylor Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No